CLINICAL TRIAL: NCT02538679
Title: A Comparison of Ultrasound Guided Transversus Abdominis Plane Nerve Block Technique Versus Laparoscopic Transversus Abdominis Plane Nerve Block Technique Versus No Block on Postoperative Opioid Consumption After Major Colorectal Surgery
Brief Title: A Comparison of Ultrasound Guided Transversus Abdominis Plane Nerve Block Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karen Zaghiyan, Clinical Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00037604
Record Dates: First submitted 2015-08-20; First posted 2015-09-02 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease; Postoperative Pain
Keywords: transversus abdominis plane block; tap block; regional anesthesia; colorectal surgery
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Pain, Postoperative | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- PLACEBO (Placebo Comparator): No TAP block performed
  Interventions: Other: Placebo
- US TAP Bupivacaine/Epinephrine (Experimental): Ultrasound guided bupivacaine 0.25% with epinephrine 1:400k will be injected to the transversus abdominis plane.
  Interventions: Drug: US TAP Bupivacaine/Epinephrine
- Lap TAP Bupivacaine/Epinephrine (Experimental): Laparoscopic guided bupivacaine 0.25% with epinephrine 1:400k will be injected to the transversus abdominis plane.
  Interventions: Drug: Lap TAP Bupivacaine/Epinephrine

INTERVENTIONS:
Other: Placebo — The usual intraoperative and postoperative pain control; NO TAP block performed
  Arms: PLACEBO
Drug: US TAP Bupivacaine/Epinephrine — Ultrasound guided bupivacaine 0.25% with epinephrine 1:400k will be injected to the transversus abdominis plane.
  Arms: US TAP Bupivacaine/Epinephrine
Drug: Lap TAP Bupivacaine/Epinephrine — Laparoscopic guided bupivacaine 0.25% with epinephrine 1:400k will be injected to the transversus abdominis plane.
  Arms: Lap TAP Bupivacaine/Epinephrine

SUMMARY:
Postoperative pain can pose significant challenges in the postoperative recovery of patients undergoing major colorectal surgery. Traditionally, opioids have played an important role in treating postoperative pain. It is well established that opioids are highly effective in relieving pain; however opioids are associated with numerous side effects that include nausea, vomiting, constipation, ileus, bladder dysfunction, respiratory depression, pruritus, drowsiness, sedation, and allergic reaction. These opioid side effects, which range in severity, can significantly interfere with discharge home following colorectal surgery. Significant interest exists in the use of local anesthetic based regional anesthesia techniques as a means to extend the analgesic window for patients undergoing colorectal surgery. Specifically, the use of the transversus abdominis plane (TAP) block as an adjunct in postoperative pain control has been widely reported in the anesthesia and colorectal surgery literature. Historically, the block was performed in a blind fashion with relative success and presently the block is typically performed either with ultrasound guidance or laparoscopic visualization. While TAP block has shown to be effective in post-operative pain control, the techniques used to place the block have not formally been compared.

The investigators are purposing a prospective, patient-blinded, randomized study of patients undergoing major colorectal surgery to compare TAP block under ultrasound guidance versus laparoscopic visualization versus no TAP block. The investigators hypothesize that laparoscopic-guided TAP block is non-inferior to ultrasound-guided TAP block with respect to perioperative pain control and either technique is superior to no TAP. In addition the investigators will measure procedural time, any adverse events related to the block, overall postoperative analgesic requirement, analgesic duration, postoperative pain scores, length of postoperative hospital stay, incidence of postoperative ileus, and overall patient satisfaction between the three groups.

DETAILED DESCRIPTION:
The proposed study is a patient-blinded, prospective randomized study to compare ultrasound-guided block of the TAP versus laparoscopic-guided TAP block versus no TAP block in patients undergoing major colorectal surgery. The primary outcome measure is analgesic requirement in morphine equivalents in the first 24 hours after surgery. Secondary outcome measures include overall postoperative analgesic requirement, postoperative pain scores, length of postoperative hospital stay, any adverse events related to TAP block, overall perioperative complications in the 30-day postoperative period and overall patient satisfaction after major colorectal surgery.

All groups will receive general anesthesia as the primary mode of anesthesia. Patients randomized to one of two treatment arms will also undergo either ultrasound-guided or laparoscopic-guided TAP block in the operating room at the conclusion of the procedure. Patients randomized to no TAP will not have a TAP block performed but will receive all routine intraoperative and postoperative analgesia as deemed appropriate by the anesthesia and primary surgical team. A standardized preoperative non-opioid pain regimen will be utilized. In the recovery room, short acting opioids for breakthrough pain will be available. Opioids will also be administered for rescue if need be. All patients will receive postoperative intravenous narcotics via patient controlled analgesia (PCA) device.

STUDY METHODS

I. Recruitment

1. Patients of the investigators will be recruited for this study during their preoperative outpatient appointments approximately one week before surgery. The study material packet containing the HIPAA and the informed consent form will be emailed to the patient for review. Thus the patient will have adequate time to ask questions and consider the study prior to scheduled surgery.
2. The patients will be contacted by one of the study investigators the morning of surgery at which time a signed consent will be obtained.
3. Only patients who have provided their written consent and indicated that they have been introduced to the study prior to meeting with the anesthesiologists on the day of surgery will be able to participate.
4. Screening procedures will make sure patients meet all inclusion criteria.

II. In the preoperative holding area:

1. An anesthesia investigator assigned to the specific case will assess patients and perform a pre-operative anesthesia assessment as per standard protocol at Cedars Sinai Medical Center (CSMC). None of this data will be recorded until written informed consent is obtained.
2. Patients will provide a detailed medical history including demographic information (e.g., age, weight, height, ethnic origin, smoking history, history of motion sickness, history of postoperative nausea and vomiting, as well as chronic analgesic usage). None of this data will be recorded until written informed consent is obtained.
3. Written informed consent will be obtained by one of the investigators.
4. Patients will be randomized in a blinded fashion by study staff to one of the groups via online randomization site, sealedenvelope.com, in a 2:2:1 fashion.

Group 1 n=100 Ultrasound guided TAP Block Group 2 n=100 Laparoscopic guided TAP Block Group 3 n=40 No TAP

III. During the intraoperative period

1. Standard anesthesia monitors will be applied: automatic blood pressure cuff, three-lead electrocardiography, capnography, and pulse oximetry will be used continuously.
2. Induction of general gnesthesia will be with propofol 2-3 mg/kg & a non-depolarizing muscle relaxant (choice will be operator dependent). Maintenance of anesthesia will be with an inhalational anesthetic.
3. The study staff performing randomization will instruct the anesthesiologist or surgeon to either block the transversus abdominis plane with ultrasound, laparoscopy, or no block.
4. For the block, a standard weight based dose (bupivacaine 0.25% with epinephrine 1:200,000, at a 1ml/kg dose) will be used for both ultrasound-guided or laparoscopic-guided block.
5. The block is administered between the costal margin and iliac crest in the anterior axillary line at 2 different sites on each side (4 injections total).
6. For ultrasound-guided TAP block, after the surgeons have completed their portion of the procedure, a member of the anesthesia research team will use sterile technique to prep the abdomen. The block is then placed bilaterally (at 2 different sites on each side of the abdomen) in the anterior axillary line, between the costal margin and iliac crest in the intermuscular plane between the internal oblique and transversus abdominis muscles using ultrasound guidance.
7. For laparoscopic-guided TAP block, the attending surgeon will perform the block at the conclusion of the procedure under laparoscopic guidance. Bilateral TAP block will be performed in the anterior axillary line between the costal margin and iliac crest. After the needle is passed through the skin, it is continued until 2 distinct "pops" are felt, indicating the needle pierced each of the 2 fascia layers (external oblique and internal oblique fascia). After injection of the correct plane, a smooth raised area of fluid covered by transversus abdominis muscle is seen with the laparoscope. The laparoscopic vision also assures that the preperitoneal plane is not injected and that the injection does not go intraperitoneal.
8. Dose of anesthetics, analgesics, local anesthetics, and IV fluid therapy during the operation will be recorded in the anesthesia record as per standard procedure. A copy of the sonographic image will be collected for each patient at the conclusion of the block.
9. Duration of surgery (from skin incision until closure) and anesthesia (from induction of spinal until discontinuation of the anesthetic drug) will be recorded in the anesthesia record as per standard procedure.

IV. PACU

1. Verbal rating scale (VRS) for pain will be assessed by the postanesthesia care unit (PACU) nurse upon arrival to recovery room, then every 30min interval until discharge.

   o Requirements for "rescue" analgesic medication will be recorded before discharge.
2. Any adverse events during the perioperative period will also be noted by PACU RN.

V. Following completion of surgery (post-operative):

1. Anesthesia will be discontinued at skin closure.
2. Patients will be transferred to the recovery room after emergence from sedation
3. Treatment of surgical pain prior to discharge from the recovery room: moderate-to-severe pain (VRS > 7): hydromorphone, 1-1.5 mg IV, moderate pain (VRS of 4-6): hydromorphone 0.5 - 1 mg IV., mild pain (VRS 2-3), hydromorphone 0.1-0.2 mg IV. Patient pain control medication will continue with the initial treatment medication for all subsequent rescue doses as needed until recovery room discharge.
4. Patient nausea, vomiting, or retching will be initially treated with ondansetron 4mg IV. Patients unresponsive to ondansetron will receive metoclopramide 10mg IV.
5. Patient discharge criteria from PACU will include: awake and alert, and has stable vital signs.

VI. Patient evaluation during hospital admission:

* VRS for pain assessment will be utilized to assess pain within the first 72 hours postoperatively and pain scores will be recorded in the patient chart by the nursing staff as per routine CSMC protocol. The average pain scores will be calculated for study analysis.
* VRS scores along with dose for all opioids will be recorded.
* Physical signs and symptoms related to the peripheral nerve block (residual sensory blockade) will be noted.
* Patient satisfaction with the overall technique will also be queried.

Pain evaluation recorded by nursing staff as per standard CSMC guidelines:

* At PACU every 30 minutes
* During admission: 12, 24, 48, and 72 hours postoperatively

Patient satisfaction with analgesia will be assessed at the time of hospital discharge or within 30 days postoperatively by telephone using a patient satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to sign an informed consent document
2. No allergies to anesthetic or analgesic medications
3. American Society of Anesthesia (ASA) physical status Class I - III adults of either sex
4. Aged 18-90 years

Exclusion Criteria:

1. Refusal to participate in the study
2. Age <18 or > 90 years
3. Contraindications to regional blockage including but not limited to:

   * Patient refusal to regional blockade
   * Infection at the site of needle insertion
   * Systemic infection
   * Bleeding diathesis or coagulopathy (as diagnosed by history or laboratory evaluation)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zaghiyan, MD, Principal Investigator — Cedars-Sinai Medical Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PLACEBO | US TAP Bupivacaine/Epinephrine | Lap TAP Bupivacaine/Epinephrine
Started | 24 | 54 | 49
Completed | 21 | 45 | 41
Not Completed | 3 | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | US TAP Bupivacaine/Epinephrine | Lap TAP Bupivacaine/Epinephrine | Total
Number analyzed (Participants) | 21 | 45 | 41 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (18.5) | 54 (16.6) | 48.4 (18.8) | 50.2 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 23 | 25 | 57
  Male | 12 | 22 | 16 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 3 | 9
  Black or African American | 3 | 5 | 6 | 14
  White | 13 | 30 | 25 | 68
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
American Society of Anesthesiologist Classification [Count of Participants; unit: Participants] — American Society of Anesthesiologist Classification grading performed by anesthesiologist prior to surgery
  Grading per standard ASA guidelines:
  ASA class I - normal healthy adult ASA class II - patients with mild systemic disease ASA class III - patients with severe systemic disease ASA class IV - patients with severe systemic disease that is a constant threat to life ASA class V - a moribund patient that is not expected to survive
  Participants
    ASA I/II | 12 | 28 | 34 | 74
    ASA III or higher | 9 | 17 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Morphine Requirement
Description: Compare ultrasound-guided block of the transversus abdominis plane (TAP) vs laparoscopic-guided TAP block, versus no TAP block on opioid consumption in the first 24 hours. Patients hospital chart was queried for use of any intravenous opioid in the first 24 hours after surgery including fentanyl or hydromorphone and conversion to morphine per standard opioid dose conversion. Total morphine equivalents then summed for the 24 hour postoperative period and compared between groups.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | PLACEBO | US TAP Bupivacaine/Epinephrine | Lap TAP Bupivacaine/Epinephrine
Number analyzed (Participants) | 21 | 45 | 41
mg | 31.4 (19.2) | 39 (35.5) | 22.8 (21.3)

ADVERSE EVENTS:
Time Frame: adverse events were recorded for the 30 day postoperative window
Arm/Group | PLACEBO | US TAP Bupivacaine/Epinephrine | Lap TAP Bupivacaine/Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/45 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/45 | 0/41
Other Adverse Events (participants affected / at risk) | 8/21 | 17/45 | 15/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=21) | US TAP Bupivacaine/Epinephrine (N=45) | Lap TAP Bupivacaine/Epinephrine (N=41)
Ileus (Gastrointestinal disorders) | 6 (6) | 11 (11) | 10 (10)
Other non-GI adverse events (Surgical and medical procedures) | 2 | 6 | 5 — any infectious, hematologic, cardiopulmonary, genitourinary, or musculoskeletal adverse events occurring in the 30 day postoperative period, monitored and recorded without regard to specific AE term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT02538679/Prot_SAP_000.pdf